CLINICAL TRIAL: NCT07391904
Title: Patient-centered Precision Medicine Lab Result Communication for Older Adults - User Experience Testing
Brief Title: Patient-centered Precision Medicine Lab Result Communication for Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Johns Hopkins University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Catherine A. Sarkisian, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-25-0471-AM-003; P30AG073104 (NIH)
Record Dates: First submitted 2026-01-22; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease (CKD); Health Communication; Patient Comprehension
Keywords: chronic kidney disease; lab result communication; Electronic Health Records; Patient Comprehension; Predictive Modeling
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of the four arms:
  Arm 1: Outcome Expectancy Condition Arm 2: Normalized Condition Arm 3: Combined Condition (Outcome Expectancy + Normalized) Arm 4: Control (current standard communication)
Masking Description: Patient participants will not be informed which version of the CKD lab result communication tool represents the newly designed version and which represents the control version.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Outcome Expectancy Condition (Experimental): Participants in this arm will first be shown a new user interface template report for communication Chronic Kidney Disease (CKD) lab results. This version emphasizes functional interpretation of kidney health and likelihood of progression over the next two years. They will answer a series of questions assessing understanding, emotional response, and likelihood of behavior change based on this presentation. Their responses will be locked in. Immediately afterward, participants will be shown the control version and asked to re-evaluate their responses with reference to their earlier answers.
  Interventions: Behavioral: Chronic Kidney Disease (CKD) Lab Result Communication Tool
- Normalization Condition (Experimental): Participants in this arm will first be shown a new user interface template report for communication CKD lab results. This version emphasizes comparative normalization by presenting personalized CKD risk in relation to results commonly observed among similar adults of comparable age and clinical characteristics. They will answer a series of questions assessing understanding, emotional response, and likelihood of behavior change based on this presentation. Their responses will be locked in. Immediately afterward, participants will be shown the control version and asked to re-evaluate their responses with reference to their earlier answers.
  Interventions: Behavioral: Chronic Kidney Disease (CKD) Lab Result Communication Tool
- Combined Condition (Outcome Expectancy + Normalization) (Experimental): Participants in this arm will first be shown a new user interface template report for communication CKD lab results. This version integrates both outcome expectancy and comparative normalization by presenting personalized CKD risk alongside functional interpretation of kidney health and contextual comparison of similar adults. They will answer a series of questions assessing understanding, emotional response, and likelihood of behavior change based on this presentation. Their responses will be locked in. Immediately afterward, participants will be shown the control version and asked to re-evaluate their responses with reference to their earlier answers.
  Interventions: Behavioral: Chronic Kidney Disease (CKD) Lab Result Communication Tool
- Control (No Intervention): Participants in this arm will only be shown control version, the standard communication CKD lab results. They will answer a series of questions assessing understanding, emotional response, and likelihood of behavior change based on this presentation.

INTERVENTIONS:
Behavioral: Chronic Kidney Disease (CKD) Lab Result Communication Tool — A behavioral intervention delivered through a personalized Electronic Health Record (EHR)-integrated lab result communication tool designed to improve emotional and cognitive responses to lab results among adults aged 65+. The tool applies behavioral science principles such as risk personalization, simplified messaging, and visual framing to reduce patient anxiety, enhance understanding, and support informed decision-making.
  Arms: Combined Condition (Outcome Expectancy + Normalization); Normalization Condition; Outcome Expectancy Condition

SUMMARY:
For adults ≥65 years and their providers, the investigators will test the usability and design of a tool to replace standard uniform reporting of lab results to patients and their providers with a new personalized Electronic Health Record (EHR) lab result communication tool that: 1) extracts patient-level data from the EHR; 2) calculates individual risk; and 3) for patients with very low risk, communicates the individualized risk information. The investigators will employ a range of User Experience (UX) research methods to understand how patient and provider users interact with the new lab result communication tool and to assess their comprehension of the lab results. This study will be conducted with both patient and provider participants. The patient participant portion of this study uses a four-arm, design to evaluate three newly designed laboratory result communication template reports compared with the current standard (control) communication. The provider participant portion of this study is non-randomized; all provider participants will review all four template reports. This will include live semi-structured interviews with the participants and review of the template report(s) of the Chronic Kidney Disease (CKD) lab result communication tool. An anonymous in-person template report feedback survey will be provided to the participants to gauge their understanding of the template report(s), clarity of the information presented, and overall satisfaction with the tool. This will be a single-visit interaction with the participant in the UCLA Health geriatric or general medicine patient waiting room.

DETAILED DESCRIPTION:
At UCLA Health over 80% of all patients >65 years view their lab results through the patient portal within one day of their availability, making this a potentially very powerful way to communicate with patients (in contrast to patient portal messaging which generally has much lower rates of viewing/uptake). Currently, lab results displayed to patients and providers via the EHR include a reference range; results outside this range are printed in red and marked by a red arrow indicator ("flagged"). Though there is a disclaimer in small text at the bottom of the report explaining that "[a] test result listed as 'abnormal' may be normal for you," the header of the report prominently features a large yellow box with the text "Abnormal."

In 2023, the investigators conducted a formal community engagement studio (CES) using well-tested methods to learn more about older adults' lived experiences with communication of lab results. The CES included 11 community stakeholders representing aging and health services organizations including but not limited to the LA County Aging and Disabilities Department, the local Area Agency on Aging (AAA), AARP California, and Watts Labor Community Action Center. Results from that CES include consensus around two key conclusions: 1) older adults want more "useful information" to accompany their lab results; 2) there is tremendous enthusiasm around the idea of individualizing communication of the results of diagnostic lab tests.

For this study, the primary analysis is to compare self-report attitudes in response to behavioral-science grounded new template reports versus each other. Four arm Randomized Controlled Trial (RCT) between unique participants. The primary analyses will assess differences between each new template report and the control communication. Secondary analyses include testing the acceptability/preference of the new template reports combined versus control across participants and also a within participant analysis for the 3 arms who receive one of the new communications first followed by the control.

ELIGIBILITY:
Patient Inclusion Criteria:

* Older adults (aged ≥65 years);
* Currently have a UCLA primary care provider (PCP);
* Enrolled in the patient portal;
* English-speaking (as the language of the tool is currently only in English, and it would be impractical to have validated translations created for all of the potential variations and derivatives of the tool template reports); and
* Without dementia or other neurocognitive disease.
* Does not have End-Stage Kidney Disease (ESKD)

Provider Inclusion Criteria:

- UCLA Health providers who care for large numbers of older adults in outpatient settings.

Patient Exclusion Criteria:

* Are under the age of 65
* Do not have a UCLA PCP;
* Are not enrolled in the patient portal;
* Are not English speaking (as the tool prototypes are only in English until final verbiage is determined);
* Are diagnosed with dementia or other neurocognitive disease.
* Have ESKD

Provider Exclusion:

- Do not care for large numbers of older adults in outpatient settings

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Compare self-report attitudes in response to behavioral-science grounded new template reports versus each other. Four arm Randomized Controlled Trial (RCT) between unique participants. | 12 months
  Participants will complete a structured post-session anonymous survey using a 4-point Likert scale titled "Emotional Response to Lab Results".
  The survey will assess emotional response and will be measured using a 4-point Likert-scale:
  1. Anxiety - A higher score indicates extremely anxious
  2. Understanding of Information - A higher score indicates understanding completely
  3. Trust - A higher score indicates trust completely
  4. Urgency - A higher score indicates extremely urgent
  5. Overall preference of new template report - A higher score indicates that the participant liked it very much.
  Responses will be compared to participants' recalled or expected emotional responses based on past experiences with standard lab result communication formats.
Providers Feedback using the new communication tool. | 12 months
  Understand how providers would feel about using the new communication tool. Document findings to support claims about preferred template report and tool effectiveness over the status quo.
  The anonymous survey will assess providers perceptions of the new designs compared with existing communication approach, including perceived improvement over the status quo, clarity of information presented, perceived preference among older adult patients, and likelihood of recommending each version for clinical use.
  Reponses will be collected using a 4-point Likert scale. The scale ranges from 1 (Strongly Disagree) to 4 (Strongly Agree).

SECONDARY OUTCOMES:
Test the acceptability of the new template reports | 12 months
  Acceptability and preference of the new template reports will be assessed among participants randomized to intervention arms 1-3. After completing the initial post-review anonymous survey of the newly designed template report, participants will additionally review the status quo lab result template report and complete a follow-up survey comparing the two versions. All patient surveys will be anonymous.
  Comparative items will assess the following:
  1. Overall preference between two designs
  2. Strength of preference - measured using a 4-point Likert-scale with a higher score indicates stronger preference
  3. Perceived clarity and ease of understanding
  4. Relative anxiety elicited by each version.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Healthy System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No